CLINICAL TRIAL: NCT01619267
Title: Device Associated Infections - Role of New Diagnostic Tools
Brief Title: Role of New Diagnostic Tool in Device (ICD / PM) Associated Infections
Acronym: DIRT
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: University Hospital Dubrava (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-008
Record Dates: First submitted 2012-06-11; First posted 2012-06-14 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Biomarkers in Device Associated Infections
Keywords: pacemaker defibrillator infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — new inflammatory biomarkers such as procalcitonine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- device associated infection: patients with proven device associated infection
- control group: patients without device associated infection

SUMMARY:
Infections related to implantable pacemakers or cardioverters defibrillators are sometimes difficult to be diagnosed. Diificulties in the diagnosis include a low sensitivity of standard markers of inflammation such as C-reactive protein or white blood cell count and the diagnosis is mainly based on the clinical presentation. The observational DIRT-study evaluates if new biomarkers may be more suitable to support a diagnosis of device associated infections than the currently available ones.

ELIGIBILITY:
Inclusion Criteria:

* device associated infections

Exclusion Criteria:

* malignancy
* cytostatic or immunomodulating therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients presenting with device associated infections
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
procalcitonine | no follow-up
  procalcitonine is determined at inclusion and correlated to infectíon status

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospital Dubrava, Zagreb, Croatia
- Germany (2):
  - Krankenhaus Landshut-Achdorf, Landshut
  - Deutsches Herzzentrum, München
- Ospedale San Pietro FBF, Rome, Italy

REFERENCES:
- [Derived] Lennerz C, Vrazic H, Haller B, Braun S, Petzold T, Ott I, Lennerz A, Michel J, Blazek P, Deisenhofer I, Whittaker P, Kolb C. Biomarker-based diagnosis of pacemaker and implantable cardioverter defibrillator pocket infections: A prospective, multicentre, case-control evaluation. PLoS One. 2017 Mar 6;12(3):e0172384. doi: 10.1371/journal.pone.0172384. eCollection 2017. PMID 28264059
- See also: Publication DIRT-Study — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0172384